CLINICAL TRIAL: NCT00521417
Title: A Randomized Controlled Study of the Efficacy of Analytic Oriented Group Psychotherapy for Psychiatric Outpatients
Brief Title: Short- and Long-term Group Psychotherapy
Acronym: KOLG-P
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oslo (Other)
Collaborators: Brigham Young University (Other)
Responsible Party: Principal Investigator, Steinar Lorentzen, professor emeritus, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aker2004-77
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Mood Disorders; Anxiety Disorders; Personality Disorders
Keywords: RCT
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Personality Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- short-term dynamic therapy (Experimental): Group therapy 20 sessions, give insight
  Interventions: Behavioral: short-term dynamic therapy
- long-term dynamic therapy (Active Comparator): Group therapy 80 sessions, give insight
  Interventions: Behavioral: long-term dynamic therapy

INTERVENTIONS:
Behavioral: short-term dynamic therapy
  Arms: short-term dynamic therapy
Behavioral: long-term dynamic therapy
  Arms: long-term dynamic therapy

SUMMARY:
A primary goal of this study is to investigate the significance of treatment duration, by comparing change after group psychotherapy of varying lengths. A secondary goal is to investigate the predictive value of selected patient variables on outcome: personality pathology, quality of object relations, presence of personality disorder, degree of initial disturbance, and education. One hundred and twenty patients from 5-6 different study sites (consisting of one coordinator and 3 therapists) will be included. Exclusion criteria are psychosis, substance abuse, and organically based symptoms. Patients are interviewed before treatment and one year after termination, and self-rated outcome measures are filled in at 3-month intervals during treatment and at termination. After an initial evaluation, patients are randomized to one of two manualized psychodynamic group psychotherapies with different treatment lengths (20 and 80 sessions). Each therapist will conduct both a short- and a long-term group, and sessions are taped in order to check treatment integrity.

DETAILED DESCRIPTION:
The primary goal is to study the effect of treatment duration, by comparing potential change during and after psychodynamic group psychotherapy of varying length (20 and 80 sessions), on measures of symptomatic distress, interpersonal problems, psychosocial functioning, and dynamic personality structure. Hypotheses related to the primary goal: Patients in short- and long-term therapy will symptomatically (SCL-90-R; Derogatis, 1977) be improved to an equal degree, while patients in long-term group psychotherapy will have a larger improvement in interpersonal problems (IIP-64; Alden et al, 1990), psychosocial functioning, and dynamic personality structure.

A secondary goal is to investigate the predictive value of selected patient variables (moderators):

• Personality pathology: Internal object relationships (QOR; Høglend et al, 2003): Patients with better object relationships will improve more both in short- and long-term therapy, and patients with poorer object relationships will improve more in long-term therapy and less in short-term therapy.

Personality disorder: Patients without personality disorders improve equally well in short- and long-term group psychotherapy, while patients with personality disorders will have a substantial reduction in criteria for personality disorder after long-term group psychotherapy.

• Severity of initial disturbance: Patients who have a high severity of the initial disturbance will do better in long-term than in short-term therapy. Patients with low severity of initial disturbance will do equally well in short- and long-term group psychotherapy.

• Education: Years of formal education (as an expression of a positive mental capacity) is included as a potential important moderator based on instructional and organizational research.

A tertiary goal is to study mediators, or mechanisms of change: Attributional Style Questionnaire (Seligman et al., 1979), Self-understanding (Mary Beth Conolly Gibbons, 2004), and Therapist Introject (Arnold, Farber, & Geller, 2004) are our primary mediators. The Therapist Introject is modified to be a 'Group Introject' measure, since experience from group psychotherapy shows that patients often internalize parts of or the-group-as-a-whole in successful therapies.

A fourth goal is to study the impact of different process variables. Studies in short-term therapy, indicate that the development of an early strong therapeutic alliance is related to a positive therapy process and outcome. This may be different on long-term therapy, where work with character defenses in the mid-phase of therapy, may lead to variations in the alliance. However, this has hardly been studied at all. A few studies of short-term group psychotherapy indicate a positive relation between cohesion and outcome, while there is a lack of similar studies of long-term therapies. The Group climate Questionnaire (GCQ) contains three subscales (engagement, avoidance and conflict), tapping degree of engagement in psychological work, reluctance to take responsibility for psychological change, and friction between members, respectively. It has been used in studies of group development, stages, and outcome, mostly in short-term groups. Again, there is a lack of studies of long-term groups. We want to compare the potentially differential development and influence of these dimensions in short- and long-term group psychotherapy.

Material and Methods

This is a randomized clinical study fulfilling the following criteria:

Patients from clinical situations Representative samples Estimation of statistical power and clinical significance Control of treatment integrity (analyzing audio recordings) Experienced therapists Treatment protocols Control for therapist effect Four or more evaluations More than one rater at each time point Specified primary result variables Evaluators are blind as to treatment type Patients are blind as to which hypotheses are tested Analysis of drop outs Intention to treat analysis Moderators are specified a priori

Patients: Inclusion criteria: Patients who consult or are referred to oupatient psychiatric centers or private pratice, and who are considered suitable for ambulant psychodynamic group psychotherapy. Exclusion criteria: Active psychotic disorder, drug or alcohol dependence as main diagnosis, organically based symptoms, e.g. brain damage, autism and adult ADHD.

Sample size, calculation of statistical power: We want to detect a moderate difference in effect-size between long-term and short-term group psychotherapy, i.e. d =.50, measured with Global Assessment of Functioning (GAF: American Psychiatric Association, 1987). In our effectiveness study (Lorentzen et al., 2002) we found that post-therapy GAF standard deviation was 5.9. We consider that 3.0 GAF-points can be seen as the least improvement that is clinically significant, i.e. d = .50, during treatment. We read directly from a nomogram (Altman, 1991) that we will need a sample size of n = 120 in order to have a power .80 with a significance level of .05 (two-tailed). This means that we need 60 patients in each group.

Patient selection: The patients are recruited from four (geographical) centers, consisting of one coordinator and 2-3 therapists. The coordinators will evaluate and diagnose the patients and randomize to the two different treatment conditions. After randomization, the patients' expectations to the therapy will be noted. The groups will be closed, but if the attrition in the long-term groups is large, new patients have to be admitted. They will be included in the study if they enter the groups during the first 6 months.

Therapists, groups: Each therapist will take one short- and one long-term group, in order to eliminate "therapist noise").

Therapies: Patients will receive two different forms of psychodynamic group psychotherapy. We have developed manuals for these two therapy formats, and the therapists have been trained in these therapy forms. They include the description of a framework for psychodynamic understanding and interventions, as well as principles that will differentiate between the two formats: e.g. degree of focus, therapist activity, and handling of the termination of the therapy. Several sessions (early, midway and in the end) will be recorded and rated in order to check treatment integrity.

Evaluation: The patients are interviewed before treatment, and three years after therapy started. The interviews will be audio-recorded and include a full psychiatric record, diagnosis (SCID I og II; Spitzer et al, 1988) and psychodynamic/structural aspects. The evaluators will be blind as to the therapy of the patients. Self-rated outcome measures are filled in every three months during the treatment.

Statistics: Pre-post-follow-up change and potential differences between the two groups that are treated differently, are examined using mixed linear modelling analyses. Clinically significant change for single patients is calculated from normative values in the population and RCI (reliable change index; Jacobson, & Truax, 1991). The predictive power of different patient variables within each treatment, will be analysed with multiple regression analyses.

Scientific board We have organized a scientific board consisting of Prof. dr. med. Per Høglend, Associate Prof. dr. med. Steinar Lorentzen, both University of Oslo, Research director dr. med. Torleif Ruud, SINTEF; and Professor, PhD Michael J. Lambert, Brigham Young University, Utah. Steinar Lorentzen will be leading the research and responsible for carrying the project through. We have one research fellow, Jan Vegard Bakali, and would like one more connected to the project. Several raters will be hired later to evaluate audio recordings of therapy and evaluation sessions.

Progression We have established four study sites around Norway (Ålesund, Stavanger, Sandnes and Oslo) and trained coordinators and therapists during spring/summer 2005. The project is licensed by the Data Inspectorate and has been presented for the Regional ethical committee for medical research, which had no objections to the project.

Inclusion of patients started August 2005 and sixteen groups have started by April 2007. All patients will have been included within the end of May 2007. All patients will have ended therapy by the end of May 2009 and will have been assessed at follow-up by summer 2010. The publication process will take place in 2010-2011, but results from parts of the study may be published earlier.

Scientific significance The study will potentially contribute to increased knowledge of the efficacy of short- and long-term dynamic group psychotherapy, and the impact of treatment duration (see attached recommendation from Professor Michael J. Lambert, Brigham Young University). We will also be able to find out more about indications for short- and long-term group psychotherapy, depending on how patient characteristics predict outcome in the two therapy forms. It has been difficult to treat patients with a personality disorder in short-term therapy, while long-term psychotherapy has shown more promising results. This study will give important information about the significance of treatment length (interaction patient characteristics x treatment length).

ELIGIBILITY:
Inclusion Criteria:

* Patients who consult or are referred to oupatient psychiatric centers or private pratice, and who are considered suitable for ambulant psychodynamic group psychotherapy.

Exclusion Criteria:

* Active psychotic disorder, drug or alcohol dependence as main diagnosis, organically based symptoms, e.g. brain damage, autism and adult ADHD.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2005-08; Primary Completion 2018-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
scl-90-R, IIP-C, GAF | before and after therapy,follow-up and every 3 months during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Lorentzen, Dr. med., Study Director — Associate Professor University of Oslo
Locations (1):
- Distriktpsykiatrisk senter Helse sunnmøre, Ålesund, Ålesund, Norway

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Lorentzen S, Ruud T, Fjeldstad A, Hoglend P. Comparison of short- and long-term dynamic group psychotherapy: randomised clinical trial. Br J Psychiatry. 2013 Sep;203(3):280-7. doi: 10.1192/bjp.bp.112.113688. Epub 2013 Sep 12. PMID 24029539